CLINICAL TRIAL: NCT04838249
Title: Investigation of the Effects of Testosterone and Estrogen on Eating Behavior, Metabolism, Energy Balance and Cardiovascular System in Transsexual Patients Undergoing Cross-sex Hormone Therapy
Brief Title: Effects of Cross-sex Hormone Therapy on Eating Behavior, Metabolism, Energy Balance and Cardiovascular System
Acronym: HHS
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Sascha Heinitz, Principal investigator, University of Leipzig
Other Study IDs: 023/20-ek
Record Dates: First submitted 2021-03-18; First posted 2021-04-09 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Transsexualism; Transgenderism; Adiposity; Eating Behavior; Arterial Stiffness; Microangiopathy
Keywords: Transsexualism; Energy expenditure; Energy balance; Eating behavior; Adiposity; Cardiovascular disease
MeSH Terms: conditions — Transsexualism; Obesity; Feeding Behavior; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Female Control: n = 20; Inclusion criteria
  informed consent, if <18 years from all legal guardians only for part B (patients will participate in all other study parts): weight stable (± 5%) for last 3 months BMI ≤ 30 kg/m² Exclusion criteria severe medical impairments (e.g., uncontrolled cardiovascular disease, severe heart failure, uncontrolled hypertension, cerebral insult, active malign disease, etc.) only for part B (patients will participate in all other study parts): Insufficiently controlled endocrine disorders Chronic pulmonary disorders Diagnosed gastrointestinal diseases History of HIV infection or ongoing chronic infection only for part D (patients will participate in all other study parts): Contraindication against performance of an MRI scan (i.e., presence of metal in body, tattoos in head/neck region, claustrophobia etc.)
- Male Control: n = 20; Inclusion criteria
  informed consent, if <18 years from all legal guardians only for part B (patients will participate in all other study parts): weight stable (± 5%) for last 3 months BMI ≤ 30 kg/m² Exclusion criteria severe medical impairments (e.g., uncontrolled cardiovascular disease, severe heart failure, uncontrolled hypertension, cerebral insult, active malign disease, etc.) only for part B (patients will participate in all other study parts): Insufficiently controlled endocrine disorders Chronic pulmonary disorders Diagnosed gastrointestinal diseases History of HIV infection or ongoing chronic infection only for part D (patients will participate in all other study parts): Contraindication against performance of an MRI scan (i.e., presence of metal in body, tattoos in head/neck region, claustrophobia etc.)
- Female cross-sex hormone therapy: n = 20; Inclusion criteria
  transsexual patients undergoing cross-sex hormone therapy informed consent, if <18 years from all legal guardians only for part B (patients will participate in all other study parts): weight stable (± 5%) for last 3 months BMI ≤ 30 kg/m²
  Exclusion criteria
  severe medical impairments (e.g., uncontrolled cardiovascular disease, etc.) self-initiated cross-sex hormone therapy before study start only for part B (patients will participate in all other study parts): Insufficiently controlled endocrine disorders Chronic pulmonary disorders Diagnosed gastrointestinal diseases History of HIV infection or ongoing chronic infection only for part D (patients will participate in all other study parts): Contraindication against performance of an MRI scan
- Male cross-sex hormone therapy: n = 20; Inclusion criteria
  transsexual patients undergoing cross-sex hormone therapy informed consent, if <18 years from all legal guardians only for part B (patients will participate in all other study parts): weight stable (± 5%) for last 3 months BMI ≤ 30 kg/m²
  Exclusion criteria
  severe medical impairments (e.g., uncontrolled cardiovascular disease, etc.) self-initiated cross-sex hormone therapy before study start only for part B (patients will participate in all other study parts): Insufficiently controlled endocrine disorders Chronic pulmonary disorders Diagnosed gastrointestinal diseases History of HIV infection or ongoing chronic infection only for part D (patients will participate in all other study parts): Contraindication against performance of an MRI scan

SUMMARY:
Current study aims to characterize five highly interconnected physiological systems in patients undergoing cross-sex hormone therapy - namely glucose and lipid metabolism, energy balance, eating behavior, functional brain networks involved in the regulation of eating behavior and the cardiovascular system - to gain novel insights into the effects of sex hormones on the human body. Gathered information will help to identify pathophysiological mechanisms for the development of overeating/obesity, insulin resistance, and cardiovascular disease. Secondarily, the relationships between the gut and oral microbiomes and metabolomes and circulating bacterial signatures will be investigated in relation to the other pervasive physiological systems.

Current study is an observational study. The decision if the patient's request for cross-sex hormone therapy can complied with (i.e., if cross-sex hormone therapy is medically indicated) is made prior to the first contact with the study center and with the outpatients clinic for Endocrinology at the University Hospital in Leipzig. Decision ifor treatment is made according to national and international guidelines. Treatment of study participants with testosterone and estradiol/antiandrogens is not affected by the study. During the course of the study no invasive interventions are being performed.

DETAILED DESCRIPTION:
1. Introduction 1.1. Transsexualism Transsexualism is a condition in which an individual's gender identity is incongruent with the assigned sex at birth. Many transsexuals suffer from severe psychological problems caused by this this incongruence, referred to as gender dysphoria. Supporting transsexuals in living in the sex with which they identify leads to amelioration of psychological problems and medical problems. In sex reassignment therapy, cross-sex hormone therapy is an essential element.

   1.2. Cross-sex hormone therapy in transsexual patients In many patients, cross sex hormone therapy is used to conduct sex change. In transmen (biological women with perceived male sex), testosterone is used for gender reassignment. In transwomen (biological men with perceived female sex), the most commonly used medication is estrogen. Successful therapy leads to the development of typical secondary sex characteristics. Data and knowledge regarding the effects of cross-sex hormone therapy on the human body, additionally to the desired sex affirming changes, is scarce.

   1.3. Investigation of the effects of estrogen and testosterone on the human body Investigating the effects of cross-sex hormone therapy provides further information on the effects of testosterone and estradiol on the human body. One of the most recognized differences between men and women regarding health is the increased cardiovascular risk of men as compared to women. In transmen, testosterone therapy leads to an increased risk for myocardial infarction. Data from the diabetes prevention program suggest that in males the probability of developing diabetes mellitus type 2, a major risk factor for cardiovascular disease is positively correlated with serum concentrations of estradiol and negatively correlated with concentrations of testosterone. Furthermore, previous studies pointed to differences in the regulation of eating behavior of men and women potentially contributing to the development of obesity and type-2-diabetes.

   Moreover, while the microbiota, known to affect host homeostasis, immunity, and metabolism, shows sex-related variations, the impact of sex hormones and gender transition on the different microbiome niches and related metabolic processes, remains largely unexplored.

   The above mentioned findings are just examples of plentiful dissimilarities in health and disease of the two sexes with unknown causes. To date studies assessing e.g. markers of cardiometabolic disease in cross-sex hormone therapy remain inconclusive.

   1.4. Purpose of this study To gain novel insights into the effects of sex hormones on the human body, current study aims to characterize four highly interconnected physiological systems in patients undergoing cross-sex hormone therapy: glucose and lipid metabolism, energy balance, eating behavior, and the cardiovascular system as well as several microbiome niches. Gathered knowledge will help to identify pathophysiological mechanisms for the development of overeating/obesity, insulin resistance, and cardiovascular disease.
2. Aims The study is designed to investigate the effects of testosterone and estradiol/cyproteron acetate in patients with gender dysphoria/transsexualism undergoing cross-sex hormone therapy in comparison to a control group without hormone therapy.

   Effects of cross-sex hormone therapy on:

   Part A Glucose and lipid metabolism Part B Body composition and energy balance control, microbiome Part C Psychobehavioral traits with a focus on eating behavior Part D (Cardio-) Vascular system

   To best possibly attribute observed effects to the applied sex hormones, baseline measurements before starting cross-sex hormone treatment will be performed (V0). Measurements will be repeated at five time points during ongoing cross sex hormone treatment (V1-5):

   V0 Baseline assessment before start of cross-sex hormone therapy V1 Three months after start of cross-sex hormone therapy V2 Six months after start of cross-sex hormone therapy V3 Twelve months after start of cross-sex hormone therapy V4 Two years after start of cross-sex hormone therapy V5 Five years after start of cross-sex hormone therapy To be able to exclude unspecific order effects of the measurements and to be able to compare obtained results with non-transsexual persons, controls not undergoing cross-sex hormone therapy matched for age, body mass index, health status (morbidity) and education will be included.
3. Research Design and Methods 3.1. Participants and recruitment This is a five year observational, non-invasive study to evaluate the effect of cross-sex hormone therapy on metabolism, eating behavior, body composition, energy expenditure, oral and the gut microbiomes, and the cardiovascular system. Results will be compared longitudinally on an intra-individual level, as well as on an inter-individual level by comparing transmen with transwomen and both groups with non-treated controls. Transsexual patients will be recruited at the outpatient clinic for Endocrinology at the University Hospital Leipzig. Patients seeking cross-sex hormone therapy will be asked before starting cross-sex hormone therapy for their willingness to participate in the study. Patients willing to participate will be screened for study eligibility. Eligible subjects will be informed about the study procedures and possible risks. Upon receiving written informed consent, the patient will be included into the study. Willingness to participate in the study will not influence the medical treatment.

A control group of men and women matched for age, body mass index, health status (morbidity) and education who are not undergoing cross-sex hormone therapy will be recruited via online advertisements.

3.2. Study procedures Seven days prior to baseline assessment, accelerometers will be handed to participants to measure physical activity. Four days prior to baseline, participants will be asked to complete a 96h activity log to objectify physical activity. Food intake will be self-assessed four days prior to baseline assessment via questionnaire as instructed by a trained dietitian. Dietary restraints will be assessed (e.g., lactose intolerance, etc.) to adjust procedures of ad libitum food intake measurement to individual needs. A tour of our metabolic unit and the MRI facilities will be given to participants and procedures explained. Subjects will be asked to fill out behavioral questionnaires at home, within one hour of completing their breakfast, to decrease variability of answers. Participants will use provided kits to collect stool samples for the gut microbiome analysis.

On the day of baseline assessment, prior to initiation of cross-sex hormone therapy/no therapy, current medical history including current medication, a physical exam including measurement of weight, waist and hip circumferences, blood pressure and heart rate will be performed. In the fasted state, blood will be drawn to measure fasting glucose, HbA1c%, serum insulin, triglycerides, total-, low- and high-density-lipoprotein concentrations. Insulin sensitivity and HOMA-IR will be calculated. The fasting blood draw will further include measurement of 17β-estradiol, progesterone, testosterone, sex-hormone binding globulin (SHBG), blood cell count, creatinine, ALAT, ASAT, GGT, TSH, and FGF21. Saliva samples will be collected in a fasted state for analysis of oral microbiome. All samples will be stored at -80 °C and then sent for commercial sequencing and metabolome analysis. In control women and transmen we will record whether menstrual cycle still persists. From each blood draw, serum will be stored at -80°C for future analyses. In order of procedures performed during baseline assessment, subjects will receive:

* Assessment of body composition: Fat mass and fat-free mass will be assessed using body impedance analysis (BIA).
* Measurement of resting energy expenditure: Baseline indirect calorimetry using a ventilated hood method will be performed in the fasted state resting energy expenditure (REE) prior to hormone substitution therapy/no therapy. The measurement will take 30 min. In brief, a clear plastic hood will be placed over the participants head with a soft collar around the neck to prevent any air leaks. The hood will be securely ventilated with room air and over 30 min. constant fractions of gases flowing out of the hood will be analyzed for carbon dioxide and oxygen concentrations. Via measurement of the respiratory quotient, calorimetric measurements will be performed during 5 min. intervals and over a period of 30 min. the subject's mean REE will be estimated. Using the ventilated hood method, adverse events are scarce and may include claustrophobia. Thus, subjects suffering from claustrophobia will be exempt from this measurement.
* Ultrasound of vessels and microperfusion: Ultrasound will be conducted to evaluate arterial stiffening (abdominal aorta and carotid artery; regional aortic strain and aortic impedance characteristics via LVOT doppler and aortic tonometry, GE Healthcare, Vivid E9 system). Peripheral near-infrared spectroscopy combined with a vascular occlusion test will be used to evaluate microperfusion (near-infrared spectroscopy, Diaspective Vision, Tivita tissue).
* Ad libitum food intake: For breakfast, subjects will undergo an ad libitum food intake situation in which they will be exposed to a buffet and asked to eat as much as they want. The buffet addresses individual dietary retrains (e.g., vegan diet). Caloric and macronutrient intake will be measured. Prior to and immediately after the buffet, participants will rate their mood, hunger, and desire to eat on a 10 cm visual analogue scale.
* Snack Food Taste Test: For assessment of taste preferences and as an additional measure of ad libitum food intake a snack food taste test will be performed. This test will be administered within 30 min. after lunch. This will be a taste test where participants will be asked to rate four types of food that will be placed in front of them in large bowls: potato chips (70 g), peanuts (100 g), Oreo cookies (100 g), and M&M's (100 g). Participants will be asked to provide mood and appetite ratings. They will then be instructed to consume as much or as little as they wish and to judge the taste of the food products using the provided rating scales. The experimenter will then leave the room and return 10 min. later, remove the bowls of food and administer a final rating scale of mood and appetite. The bowls of food will be weighed before and after the taste test as a measure of food and calorie intake.
* Response to thermic stimuli: Via an electrode positioned below the base of the index finger (C6) of the participant's non-dominant hand, thermic stimuli (cold versus warm) will be administered and subjects will be asked to indicate cold/warmth perception. Perception of cold will be measured four times in a row, followed by warmth perception. Then thermal discomfort will be triggered via administration of one cold versus one warm stimulus.
* Measurement of taste perception and smell: Administration of standardized gustatory and olfactory stimuli will enable the assessment of (non)specific taste perception and the subject's ability to perceive certain scents. Taste perception will be assessed one at a time by placing paper slip on the participant's tongue that had been coated with one specific, known flavor. Similarly, the participant's ability to perceive certain scents will be tested. In this case, specific, known scents will be placed in front of the nose of the participant who will be asked to determine the scent and then asked to rate it.
* Sex hormone deposition in hair: Using liquid chromatography-mass spectrometry, deposition of sex hormones in hair will be measured (time points V2-V4). For this purpose, a small amount of hair will be removed from the occipital region of the subject's head and then analyzed.
* Gut, oral microbiome, circulating bacterial signature in the blood and metabolomics: Participants in the study will collect stool samples at home using a provided kit and bring them to the study visit. This kit includes a disposable tray and vials for metagenome sequencing. Additionally, saliva samples will be collected at the study center after fasting, along with blood for microbiome and metabolome analyses. Gut microbiome and oral microbiome will be sent for commercial library preparation and sequencing of whole genome metagenomics. Bacterial DNA in the blood will be analyzed using 16S rRNA Amplicon sequencing and stool, oral and circulating metabolomes will be subjected to commercial metabolomics via gas liquid chromatography-mass spectrometry (GLC-MS).
* Visit to our clinical outpatient unit (transgender subjects only): Based on our unit-specific standards of care, subjects will receive a prescription for hormones intended to induce transformation to the other sex (cyproterone acetate + testosterone/estradiol) and advised to begin administration of their first dose of medication on day 1 of our study. Patients will be advised to continue with treatment according to our unit-specific standards of care for subjects with gender dysphoria undergoing hormone substitution therapy.

Upon baseline assessment, cross-sex hormone treatment versus no treatment will commence. Study procedures for V2 through V5 are the same as the above mentioned.

ELIGIBILITY:
Inclusion Criteria:

* transsexual patients undergoing cross-sex hormone therapy versus controls
* able to give informed consent, if <18 years from all legal guardians
* only for part B (patients will participate in all other study parts): weight stable (± 5%) for last 3 months, BMI ≤ 30 kg/m2

Exclusion Criteria:

* severe medical impairments (e.g., uncontrolled cardiovascular disease, severe heart failure, uncontrolled hypertension, cerebral insult, active malign disease, etc.)
* self-initiated cross-sex hormone therapy before study start only for part B (patients will participate in all other study parts): Insufficiently controlled endocrine disorders (Cushing's disease, other uncontrolled pituitary disorders, uncontrolled hypothyroidism, hyperthyroidism, etc.)
* Chronic pulmonary disorders, including chronic obstructive pulmonary disease that would limit ability to follow the protocol (investigator judgment) and obstructive sleep apnea syndrome; only subjects with mild or exercise-induced asthma on no medications or on beta-adrenergic agonists only will be allowed to enter the study (provided use of these agents is not required for 1 week before
* Diagnosed gastrointestinal diseases, including inflammatory bowel diseases (e.g. Crohn's disease and ulcerative colitis), malabsorption syndromes (e.g. celiac disease), gastric ulcer (active); only subjects with gastro-esophageal reflux will be allowed to enter the study entry).
* History of HIV infection or ongoing chronic infection (such as tuberculosis)
* only for part D (patients will participate in all other study parts): Contraindication against performance of an MRI scan (i.e., presence of metal in body, tattoos in head/neck region, claustrophobia etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transsexual patients will be recruited in the outpatient clinic for Endocrinology at the University Hospital Leipzig. Patients seeking cross-sex hormone therapy will be asked before starting cross-sex hormone therapy for their willingness to participate in the study. If the patients would like to participate, a screening of in- and exclusion criteria will be performed. If the patient matches the criteria, the patient will be informed about the study procedures and eventual risks and if written consent will be given, the patient will be included into the study. Willingness to participate in the study will not influence the medical treatment. A control group of men and women matched for age, body mass index, health status and education who are nor undergoing cross-sex hormone therapy will be recruited through advertisements in the internet.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure | up to one year
  To examine short-term and longer-term effects of cross-sex hormone therapy on changes in resting energy expenditure (kcal/d).
Vascular stiffness | up to five years
  To examine short-term and longer-term effects of cross-sex hormone therapy on changes in vascular stiffness (change from baseline using cm/s to assess arterial stiffness).
Insulin sensitivity | up to five years
  To examine short-term and longer-term effects of cross-sex hormone therapy on changes in insulin sensitivity (change from baseline using HOMA-IR to assess insulin sensitivity).
Food intake | up to one year
  To examine short-term and longer-term effects of cross-sex hormone therapy on changes ad libitum food intake (change from baseline in kcal).
Weight change | up to one year
  To examine short-term and longer-term effects of cross-sex hormone therapy on weight change (change from baseline in kg).

SECONDARY OUTCOMES:
Taste perception | up to five years
  To examine short-term and longer-term effects of cross-sex hormone therapy on taste perception (change from baseline score during test assessing taste perception).
Olfaction | up to five years
  To examine short-term and longer-term effects of cross-sex hormone therapy on olfaction (change from baseline score during test assessing taste perception).
Gut, oral and circulating microbiomes and metabolomes | up to five years
  To examine short-term and longer-term effects of cross-sex hormone therapy on gut and oral microbiome composition (change of overall diversity, functional potential) as well as decompartmentalization effects on bacterial signature in the blood. These analyses will be coupled to metabolomics to delineate the metabolic outputs of the microbial niches and relate this system to the other studied physiological systems in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Blueher, MD, Study Chair — Helmholtz Institute for Metabolic, Obesity and Vascular Research
Locations (1):
- Helmholtz Institute for Metabolic, Obesity and Vascular Research, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data on primary outcomes of all study arms (A-E) will be shared upon personal and reasonable request in an anonymized manner.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Up to two years post termination of recruitment.
Access Criteria: Personal and reasonable request.

REFERENCES:
- [Background] Asarian L, Geary N. Sex differences in the physiology of eating. Am J Physiol Regul Integr Comp Physiol. 2013 Dec;305(11):R1215-67. doi: 10.1152/ajpregu.00446.2012. Epub 2013 Jul 31. PMID 23904103
- [Background] Berry C, Sidik N, Pereira AC, Ford TJ, Touyz RM, Kaski JC, Hainsworth AH. Small-Vessel Disease in the Heart and Brain: Current Knowledge, Unmet Therapeutic Need, and Future Directions. J Am Heart Assoc. 2019 Feb 5;8(3):e011104. doi: 10.1161/JAHA.118.011104. No abstract available. PMID 30712442
- [Background] Butler E, Chin M, Aneman A. Peripheral Near-Infrared Spectroscopy: Methodologic Aspects and a Systematic Review in Post-Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1407-1416. doi: 10.1053/j.jvca.2016.07.035. Epub 2016 Jul 28. No abstract available. PMID 27876185
- [Background] Coleman E, Bockting W, Botzer M, et al. (2012) Standards of Care for the Health of Transsexual, Transgender, and Gender-Nonconforming People, Version 7. International Journal of Transgenderism 13:165-232
- [Background] Coutinho T, Borlaug BA, Pellikka PA, Turner ST, Kullo IJ. Sex differences in arterial stiffness and ventricular-arterial interactions. J Am Coll Cardiol. 2013 Jan 8;61(1):96-103. doi: 10.1016/j.jacc.2012.08.997. Epub 2012 Nov 1. PMID 23122799
- [Background] Defreyne J, Van de Bruaene LDL, Rietzschel E, Van Schuylenbergh J, T'Sjoen GGR. Effects of Gender-Affirming Hormones on Lipid, Metabolic, and Cardiac Surrogate Blood Markers in Transgender Persons. Clin Chem. 2019 Jan;65(1):119-134. doi: 10.1373/clinchem.2018.288241. PMID 30602477
- [Background] Diehl JM, Staufenbiel T (2006) Inventar zum Essverhalten und Gewichtsproblemen (IEG). 4th ed. Verlag Dietmar Klotz, Eschborn, Germany
- [Background] DuPont JJ, Kenney RM, Patel AR, Jaffe IZ. Sex differences in mechanisms of arterial stiffness. Br J Pharmacol. 2019 Nov;176(21):4208-4225. doi: 10.1111/bph.14624. Epub 2019 May 11. PMID 30767200
- [Background] Erdener SE, Dalkara T. Small Vessels Are a Big Problem in Neurodegeneration and Neuroprotection. Front Neurol. 2019 Aug 16;10:889. doi: 10.3389/fneur.2019.00889. eCollection 2019. PMID 31474933
- [Background] Garner DM, Garfinkel PE. The Eating Attitudes Test: an index of the symptoms of anorexia nervosa. Psychol Med. 1979 May;9(2):273-9. doi: 10.1017/s0033291700030762. PMID 472072
- [Background] Goldman RL, Borckardt JJ, Frohman HA, O'Neil PM, Madan A, Campbell LK, Budak A, George MS. Prefrontal cortex transcranial direct current stimulation (tDCS) temporarily reduces food cravings and increases the self-reported ability to resist food in adults with frequent food craving. Appetite. 2011 Jun;56(3):741-6. doi: 10.1016/j.appet.2011.02.013. Epub 2011 Feb 23. PMID 21352881
- [Background] Horstmann A, Busse FP, Mathar D, Muller K, Lepsien J, Schlogl H, Kabisch S, Kratzsch J, Neumann J, Stumvoll M, Villringer A, Pleger B. Obesity-Related Differences between Women and Men in Brain Structure and Goal-Directed Behavior. Front Hum Neurosci. 2011 Jun 10;5:58. doi: 10.3389/fnhum.2011.00058. eCollection 2011. PMID 21713067
- [Background] Houben K. Overcoming the urge to splurge: influencing eating behavior by manipulating inhibitory control. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):384-8. doi: 10.1016/j.jbtep.2011.02.008. Epub 2011 Feb 24. PMID 21450264
- [Background] Huxley VH, Wang J. Cardiovascular sex differences influencing microvascular exchange. Cardiovasc Res. 2010 Jul 15;87(2):230-42. doi: 10.1093/cvr/cvq142. Epub 2010 May 21. PMID 20495187
- [Background] Kautzky-Willer A, Harreiter J. Sex and gender differences in therapy of type 2 diabetes. Diabetes Res Clin Pract. 2017 Sep;131:230-241. doi: 10.1016/j.diabres.2017.07.012. Epub 2017 Jul 13. PMID 28779681
- [Background] Lyle AN, Raaz U. Killing Me Unsoftly: Causes and Mechanisms of Arterial Stiffness. Arterioscler Thromb Vasc Biol. 2017 Feb;37(2):e1-e11. doi: 10.1161/ATVBAHA.116.308563. PMID 28122777
- [Background] Kim JY, Park JB, Kim DS, Kim KS, Jeong JW, Park JC, Oh BH, Chung N; KAAS investigators. Gender Difference in Arterial Stiffness in a Multicenter Cross-Sectional Study: The Korean Arterial Aging Study (KAAS). Pulse (Basel). 2014 May;2(1-4):11-7. doi: 10.1159/000365267. Epub 2014 Aug 14. PMID 26587439
- [Background] Draijer M, Hondebrink E, van Leeuwen T, Steenbergen W. Review of laser speckle contrast techniques for visualizing tissue perfusion. Lasers Med Sci. 2009 Jul;24(4):639-51. doi: 10.1007/s10103-008-0626-3. Epub 2008 Dec 3. PMID 19050826
- [Background] Meerwijk EL, Sevelius JM. Transgender Population Size in the United States: a Meta-Regression of Population-Based Probability Samples. Am J Public Health. 2017 Feb;107(2):e1-e8. doi: 10.2105/AJPH.2016.303578. PMID 28075632
- [Background] Meule A, Muller A, Gearhardt AN, Blechert J. German version of the Yale Food Addiction Scale 2.0: Prevalence and correlates of 'food addiction' in students and obese individuals. Appetite. 2017 Aug 1;115:54-61. doi: 10.1016/j.appet.2016.10.003. Epub 2016 Oct 4. PMID 27717658
- [Background] Nadort A, Kalkman K, van Leeuwen TG, Faber DJ. Quantitative blood flow velocity imaging using laser speckle flowmetry. Sci Rep. 2016 Apr 29;6:25258. doi: 10.1038/srep25258. PMID 27126250
- [Background] Nota NM, Wiepjes CM, de Blok CJM, Gooren LJG, Kreukels BPC, den Heijer M. Occurrence of Acute Cardiovascular Events in Transgender Individuals Receiving Hormone Therapy. Circulation. 2019 Mar 12;139(11):1461-1462. doi: 10.1161/CIRCULATIONAHA.118.038584. No abstract available. PMID 30776252
- [Background] Pudel V, Westhöfer J (1989) Fragebogen zum Eßverhalten (FEV). Göttingen, Toronto, Zürich, Verlag für Psychologie Dr. C. J. Hogrefe
- [Background] Puschel J, Miehle K, Muller K, Villringer A, Stumvoll M, Fasshauer M, Schlogl H. Beneficial effects of leptin substitution on impaired eating behavior in lipodystrophy are sustained beyond 150 weeks of treatment. Cytokine. 2019 Jan;113:400-404. doi: 10.1016/j.cyto.2018.10.012. Epub 2018 Oct 24. PMID 30539782
- [Background] Raaz U, Schellinger IN, Chernogubova E, Warnecke C, Kayama Y, Penov K, Hennigs JK, Salomons F, Eken S, Emrich FC, Zheng WH, Adam M, Jagger A, Nakagami F, Toh R, Toyama K, Deng A, Buerke M, Maegdefessel L, Hasenfuss G, Spin JM, Tsao PS. Transcription Factor Runx2 Promotes Aortic Fibrosis and Stiffness in Type 2 Diabetes Mellitus. Circ Res. 2015 Aug 28;117(6):513-24. doi: 10.1161/CIRCRESAHA.115.306341. Epub 2015 Jul 24. PMID 26208651
- [Background] Raaz U, Zollner AM, Schellinger IN, Toh R, Nakagami F, Brandt M, Emrich FC, Kayama Y, Eken S, Adam M, Maegdefessel L, Hertel T, Deng A, Jagger A, Buerke M, Dalman RL, Spin JM, Kuhl E, Tsao PS. Segmental aortic stiffening contributes to experimental abdominal aortic aneurysm development. Circulation. 2015 May 19;131(20):1783-95. doi: 10.1161/CIRCULATIONAHA.114.012377. Epub 2015 Apr 22. PMID 25904646
- [Background] Ruaro B, Smith V, Sulli A, Decuman S, Pizzorni C, Cutolo M. Methods for the morphological and functional evaluation of microvascular damage in systemic sclerosis. Korean J Intern Med. 2015 Jan;30(1):1-5. doi: 10.3904/kjim.2015.30.1.1. Epub 2014 Dec 30. PMID 25589827
- [Background] S3-Leitlinie zur Diagnostik, Beratung und Behandlung: Geschlechtsinkongruenz, Geschlechtsdysphorie und Trans-Gesundheit. AWMF-Register-Nr. 138, 001. Available at https://www.awmf.org/uploads/tx_szleitlinien/138-001l_S3_Geschlechtsdysphorie-Diagnostik-Beratung-Behandlung_2019-02.pdf, accessed 3.1.2020
- [Background] Schellinger IN, Mattern K, Raaz U. The Hardest Part. Arterioscler Thromb Vasc Biol. 2019 Jul;39(7):1301-1306. doi: 10.1161/ATVBAHA.118.311578. Epub 2019 May 9. PMID 31242028
- [Background] Schlogl H, Kabisch S, Horstmann A, Lohmann G, Muller K, Lepsien J, Busse-Voigt F, Kratzsch J, Pleger B, Villringer A, Stumvoll M. Exenatide-induced reduction in energy intake is associated with increase in hypothalamic connectivity. Diabetes Care. 2013 Jul;36(7):1933-40. doi: 10.2337/dc12-1925. Epub 2013 Mar 5. PMID 23462665
- [Background] Schlogl H, Muller K, Horstmann A, Miehle K, Puschel J, Villringer A, Pleger B, Stumvoll M, Fasshauer M. Leptin Substitution in Patients With Lipodystrophy: Neural Correlates for Long-term Success in the Normalization of Eating Behavior. Diabetes. 2016 Aug;65(8):2179-86. doi: 10.2337/db15-1550. Epub 2016 May 10. PMID 27207511
- [Background] Volgman AS, Bairey Merz CN, Aggarwal NT, Bittner V, Bunch TJ, Gorelick PB, Maki P, Patel HN, Poppas A, Ruskin J, Russo AM, Waldstein SR, Wenger NK, Yaffe K, Pepine CJ. Sex Differences in Cardiovascular Disease and Cognitive Impairment: Another Health Disparity for Women? J Am Heart Assoc. 2019 Oct;8(19):e013154. doi: 10.1161/JAHA.119.013154. Epub 2019 Sep 24. No abstract available. PMID 31549581
- [Background] Wang X, Wang Y, Ma Z, Xu Y, Wu Q. Indirect calorimetry using a ventilated hood may be easier than using a facemask to achieve steady state when measuring resting energy expenditure. Nutr Res. 2017 Dec;48:33-39. doi: 10.1016/j.nutres.2017.10.010. Epub 2017 Oct 10. PMID 29246279
- [Derived] Zimmermann P, Kaar M, Bokeloh T, Moll L, Labinski F, Eippert F, Bluher M, Stumvoll M, Heinitz S, Schlogl H. Changes in temperature perception in transgender persons undergoing gender-affirming hormone therapy. Commun Med (Lond). 2026 Feb 7. doi: 10.1038/s43856-026-01420-0. Online ahead of print. PMID 41654592